CLINICAL TRIAL: NCT05513456
Title: Ethnic and Gender Based Admittance Patterns in the ICU, a Multicenter, International Randomized Survey Study
Brief Title: Ethnic and Gender Based Admittance Patterns in the ICU
Acronym: EGAP-ICU
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Max Bell, Principal Investigator, Karolinska Institutet
Other Study IDs: EGAP-ICU Project Implicit
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Critical Illness; Gender Equality; Discrimination, Sex; Discrimination, Racial
MeSH Terms: conditions — Critical Illness; Sexism; Racism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Randomization to a different factors in the case descriptions — The case descriptions will include factors like age, co-morbid status and acute physiological parameters; but the factor of sex/gender will be randomized. Moreover, randomization to case description of typical vs non-typical national name will be done.

SUMMARY:
The dominating proportion of patients in the ICU are men. Studies indicate that men receive more mechanical ventilation, vasoactive drugs, renal replacement therapy, invasive monitoring and have longer length of stay in the ICU. These differences do not unambiguously translate into a survival benefit for men; if survival would be altered if women were admitted to ICU in the same extent is unknown.

Factors affecting ICU admission include age, co-morbidities, physiological parameters (indicating severity of the acute illness) and, additionally, the number of available ICU beds. Factors that should not affect ICU admission include patient gender or ethnicity.

This study aims at studying if bias against women and people of certain ethnicities exist. Do clinicians have differing thresholds for ICU admission due to non-medical reasons?

The investigators propose testing this hypothesis using a blinded randomized factorial survey study.

DETAILED DESCRIPTION:
Background Differing treatment of men and women in several fields of health care is receiving growing attention. This includes care of the critically ill, as awareness of intensive care has dramatically increased during the last years. Critically ill patients are treated in Intensive Care Units (ICU), one of the most expensive and advanced types of care. It is therefore essential that resources are adequately used so that the patient most in need is selected for intensive care, but also that no patient in need is left without.

The dominating proportion of patients in the ICU are men. Studies indicate that men receive more mechanical ventilation, vasoactive drugs, renal replacement therapy, invasive monitoring and have longer length of stay in the ICU. It has also been shown that women and men with severe sepsis receive differential care in the emergency department. These differences do not unambiguously translate into a survival benefit for men; studies show conflicting results. One could only speculate if survival figures would be altered if women were admitted to ICU in the same extent. Sex is a biological variable that affects the immune system and changes throughout life. It is proposed that sex hormones have an impact on how the severity of an illness progresses, where female sex hormones are suggested to have a protective effect. This could partly explain male dominance in the ICU. There is no clear evidence that care given in the ICU should be tailored after the sex of the patient. Then again, there is no clear evidence that the medical care should not be tailored after the sex of the patient. Differing care provided to men and women is therefore controversial. If differences exist, it must be ruled out that it is caused by gender bias, unintentional or not.

As discussed in a recently published Guidance on Reporting of Race and Ethnicity in Medical and Science Journals, Ethnicity are social constructs, without scientific or biological meaning. However, studies including ethnicity may be useful to improve understanding and knowledge of disparities and inequities in health care. Three decades ago, US Department of Health and Human Services published a report on Black and minority health, highlighting ethnic differences. (S Department of Health and Human Services. Report of the Secretary's Task Force on Black and Minority Health. 1985. https://collections.nlm.nih.gov/catalog/nlm:nlmuid-8602912-mvset). Whilst recent studies show reductions in racial and ethnic differences in self-reported health status and health care access and affordability, variances persist. During the COVID-19 pandemic it has become apparent that differences in progression to severe disease exist. In a cohort study using the OpenSAFELY platform in England, including more than 17 million adults, some minority ethnic populations had increased risk of severe COVID-19 as compared with the White population, also after taking other factors of importance into account.

Specific aims When admitting patients to our ICUs, do clinicians discriminate against certain ethnicities? Are thresholds for admitting men lower than for women? The investigators hypothesize that differing ICU admission thresholds exist, due to non-medical reasons.

Method The investigators propose testing this hypothesis using a blinded randomized factorial survey study.

This survey will consist of multiple iterations of eight separate cases, describing a patient in the ward or in the emergency room that may need ICU admission. Co-morbid data, age, physiological parameters will be described followed by a YES/NO: would you admit this patient to your ICU, considering a "normal" ICU situation in your hospital. A count-down timer for each case will ensure that the YES/NO response comes quickly, and whilst a paper case can never mimic a real clinical situation, making fast decisions is a part of how intensivists work.

The factors affecting ICU admission are usually considered to be age, co-morbidities, physiological parameters (indicating severity of the acute illness) and, additionally, the number of available ICU beds. Factors that should not affect ICU admission include patient gender or ethnicity.

In order to test if gender and/or ethnicity affects ICU admission the survey will be randomized in several ways. Essentially, multiple different versions of the survey will exist. We will tweak the age and number of co-morbid conditions described. It is likely, but not certain, that higher patient age and more co-morbid conditions will be associated will lower admission rates. The same association is expected during a theoretical pandemic situation, with strained resources.

Unbeknown to the respondents, the cases will be randomized to describe a man or a woman. Thus, the cases can be in the order of Male, Female, M, F or reversed: F,M,F,M and so on. In one of the eight cases, the name of the patient will be a non-typical national name.

To make this generalizable and overall successful, the investigators think it is paramount to have the survey translated to French, German, Spanish and to make it simple to answer. Preferably the survey should take less than 10 minutes to complete. Moreover, sending emails, through the national organizations, might improve generalizability. Using a survey link, for instance via twitter, could create a selection bias in who chooses to click on such a link.

(This research group has done this before, so it can be done. Luckily for this project, it is not a widely cited study. https://www.nature.com/articles/s41598-019-50836-3 )

ELIGIBILITY:
Inclusion Criteria:

We will include intensive care physicians, both in training and specialists as responders in this randomized survey study

Exclusion Criteria:

We will exclude "button-mashers", i.e. participating respondents that toggle through the case descriptions faster than they possibly could read the case description. A case answered <20 seconds will be ruled out.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Intensive care physicians and other physicians working with admission (or non-admission) of critically ill patients across the world are eligible to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-05-31 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Ratio of ICU admission men vs women | Through study completion, an average of 1 year
  Exact same case descriptions except for the fact that the sex/gender is randomized
Ratio of ICU admission ethnic background | Through study completion, an average of 1 year
  Exact same case descriptions except for the fact that the name/ethnic background is randomized

SECONDARY OUTCOMES:
Time to ICU admission men vs women | Through study completion, an average of 1 year
  Do respondents take longer to decide to admit women compared to men?
Time to ICU admission ethnic background | Through study completion, an average of 1 year
  Do respondents take longer to decide to admit descriptions of patients with "other" ethnic background compared to "normal" ethnic background?
Time-out sex/gender | Through study completion, an average of 1 year
  Do respondents more often run out of time in thinking about admitting women compared to men?
Time-out described ethnicity | Through study completion, an average of 1 year
  Do respondents more often run out of time in thinking about admitting descriptions of patients with "other" ethnic background compared to "normal" ethnic background?

CONTACTS AND LOCATIONS:
Overall Officials: Max Bell, MD, PhD, Principal Investigator — Department of Physiology and Pharmacology, Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
The IPD consists of respondent country, respondent sex (M/F/other), size of hospital (university vs non-university hospital), specialist/in training, respondent age group in brackets of 10.
  It is paramount that the physicians responding to this survey know that we will not collect precise individual data, nor share the block data we do collect.

REFERENCES:
- [Background] Mahmood K, Eldeirawi K, Wahidi MM. Association of gender with outcomes in critically ill patients. Crit Care. 2012 May 22;16(3):R92. doi: 10.1186/cc11355. PMID 22617003
- [Background] Valentin A, Jordan B, Lang T, Hiesmayr M, Metnitz PG. Gender-related differences in intensive care: a multiple-center cohort study of therapeutic interventions and outcome in critically ill patients. Crit Care Med. 2003 Jul;31(7):1901-7. doi: 10.1097/01.CCM.0000069347.78151.50. PMID 12847381
- [Background] Fowler RA, Sabur N, Li P, Juurlink DN, Pinto R, Hladunewich MA, Adhikari NK, Sibbald WJ, Martin CM. Sex-and age-based differences in the delivery and outcomes of critical care. CMAJ. 2007 Dec 4;177(12):1513-9. doi: 10.1503/cmaj.071112. Epub 2007 Nov 14. PMID 18003954
- [Background] Samuelsson C, Sjoberg F, Karlstrom G, Nolin T, Walther SM. Gender differences in outcome and use of resources do exist in Swedish intensive care, but to no advantage for women of premenopausal age. Crit Care. 2015 Mar 30;19(1):129. doi: 10.1186/s13054-015-0873-1. PMID 25887421
- [Background] Sunden-Cullberg J, Nilsson A, Inghammar M. Sex-based differences in ED management of critically ill patients with sepsis: a nationwide cohort study. Intensive Care Med. 2020 Apr;46(4):727-736. doi: 10.1007/s00134-019-05910-9. Epub 2020 Jan 23. PMID 31974918
- [Background] Zettersten E, Jaderling G, Bell M, Larsson E. Sex and gender aspects on intensive care. A cohort study. J Crit Care. 2020 Feb;55:22-27. doi: 10.1016/j.jcrc.2019.09.023. Epub 2019 Oct 25. PMID 31683118
- [Background] Knoferl MW, Angele MK, Diodato MD, Schwacha MG, Ayala A, Cioffi WG, Bland KI, Chaudry IH. Female sex hormones regulate macrophage function after trauma-hemorrhage and prevent increased death rate from subsequent sepsis. Ann Surg. 2002 Jan;235(1):105-12. doi: 10.1097/00000658-200201000-00014. PMID 11753049
- [Background] Mizushima Y, Wang P, Jarrar D, Cioffi WG, Bland KI, Chaudry IH. Estradiol administration after trauma-hemorrhage improves cardiovascular and hepatocellular functions in male animals. Ann Surg. 2000 Nov;232(5):673-9. doi: 10.1097/00000658-200011000-00009. PMID 11066139
- [Background] Flanagin A, Frey T, Christiansen SL; AMA Manual of Style Committee. Updated Guidance on the Reporting of Race and Ethnicity in Medical and Science Journals. JAMA. 2021 Aug 17;326(7):621-627. doi: 10.1001/jama.2021.13304. No abstract available. PMID 34402850
- [Background] Mahajan S, Caraballo C, Lu Y, Valero-Elizondo J, Massey D, Annapureddy AR, Roy B, Riley C, Murugiah K, Onuma O, Nunez-Smith M, Forman HP, Nasir K, Herrin J, Krumholz HM. Trends in Differences in Health Status and Health Care Access and Affordability by Race and Ethnicity in the United States, 1999-2018. JAMA. 2021 Aug 17;326(7):637-648. doi: 10.1001/jama.2021.9907. PMID 34402830
- [Background] Mathur R, Rentsch CT, Morton CE, Hulme WJ, Schultze A, MacKenna B, Eggo RM, Bhaskaran K, Wong AYS, Williamson EJ, Forbes H, Wing K, McDonald HI, Bates C, Bacon S, Walker AJ, Evans D, Inglesby P, Mehrkar A, Curtis HJ, DeVito NJ, Croker R, Drysdale H, Cockburn J, Parry J, Hester F, Harper S, Douglas IJ, Tomlinson L, Evans SJW, Grieve R, Harrison D, Rowan K, Khunti K, Chaturvedi N, Smeeth L, Goldacre B; OpenSAFELY Collaborative. Ethnic differences in SARS-CoV-2 infection and COVID-19-related hospitalisation, intensive care unit admission, and death in 17 million adults in England: an observational cohort study using the OpenSAFELY platform. Lancet. 2021 May 8;397(10286):1711-1724. doi: 10.1016/S0140-6736(21)00634-6. Epub 2021 Apr 30. PMID 33939953